CLINICAL TRIAL: NCT05808920
Title: The RESCUE Study: Survival and Functional Outcomes Following Salvage Surgery for RESidual or reCurrent sqUamous cEll Carcinoma of the Head and Neck
Acronym: RESCUE
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 5752
Record Dates: First submitted 2023-02-08; First posted 2023-04-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Molecular Docking Simulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, saliva and tumour tissue samples will be collected for analysis as per the protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Participants with previous diagnosis of H&N SCC treated with radiotherapy. Recurrent, residual, or new primary SCC of the oropharynx, oral cavity, larynx, and hypopharynx treated with salvage surgery
  Interventions: Genetic: Molecular Analyses

INTERVENTIONS:
Genetic: Molecular Analyses — Nucleic acid extraction, protein analysis. Tumour tissue, blood and saliva samples collected.

SUMMARY:
The RESCUE study is a combined retrospective and prospective multicentre cohort study investigating the survival and functional outcomes in patients undergoing salvage surgery for recurrent, residual, and new primary head and neck squamous cell carcinoma (SCC).

Additionally, the RESCUE study will contain an exploratory molecular analysis of consenting patients to assess the relationship between cancer genomics, previous radiotherapy, and recurrence in head and neck cancer.

DETAILED DESCRIPTION:
The RESCUE study is a combined retrospective and prospective multicentre cohort study investigating the survival and functional outcomes in patients undergoing salvage surgery for recurrent, residual, and new primary head and neck squamous cell carcinoma (SCC).

Additionally, the RESCUE study will contain an exploratory molecular analysis of consenting patients to assess the relationship between cancer genomics, previous radiotherapy, and recurrence in head and neck cancer.

The aim of this study is to determine the survival, functional and quality of life outcomes of patients undergoing all salvage surgery for recurrent, residual and new primary head and neck SCC, and to establish the genetic architecture and clonal evolution H&N SCC after previous treatment for radiotherapy cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18
2. Previous H&N SCC treated with radiotherapy with or without chemotherapy
3. Local or regionally recurrent, residual, or new primary SCC of the oropharynx, oral cavity, larynx, and hypopharynx
4. Ability to give informed consent for biological sample collection (molecular analysis study only)

Exclusion Criteria:

1. Nasopharyngeal and cutaneous SCC of the H&N
2. Thyroid, salivary gland, and non-squamous cell H&N cancers
3. Presence of distant metastasis (M1) or surgically inoperable T4b tumours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with recurrent, residual or new primary head and neck SCC following previous treatment with radiotherapy with or without chemotherapy who have undergone or will undergo salvage surgical resection of their cancer. Head and neck subsites including the oropharynx, oral cavity, larynx and hypopharynx will be included. H&N SCC of nasopharyngeal and cutaneous origins, non-SCC, thyroid and salivary gland tumours of the head and neck will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Ascertain the 2-year disease-free survival post salvage surgery | Study duration is 3 years to include 1 year recruitment period. Active follow-up for patients is up to 2 years.
  Ascertain the 2-year disease-free survival post salvage surgery for recurrent/ residual/ new primary head and neck SCC (split cohort of prospective and retrospective patients)

SECONDARY OUTCOMES:
Define the 2- and 5-year overall and disease specific survival in retrospectively identified patients | Study duration is 3 years to include 1 year recruitment period. Active follow-up for prospective patients is up to 2 years. Follow-up for retrospective patients is up to 5 years.
  Define the 2- and 5-year overall and disease specific survival in retrospectively identified patients undergoing salvage surgery for recurrent/ residual/ new primary head and neck SCC
Define the 2 year overall and disease specific survival in prospectively identified patients | Study duration is 3 years to include 1 year recruitment period. Active follow-up for patients is up to 2 years.
  Define the 2 year overall and disease specific survival in prospectively identified patients undergoing salvage surgery for recurrent/ residual/ new primary head and neck SCC
Report on gross functional outcomes by documenting rates of gastrostomy and tracheostomy dependence at 1-year post-salvage surgery. | Study duration is 3 years with up to 2 years follow-up in prospective and up to 5 years follow-up in retrospective patients. Functional outcomes will be measured from the date of surgery.
  Report on gross functional outcomes by documenting rates of gastrostomy and tracheostomy dependence at 1-year post-salvage surgery.
For the prospective cohort assess the overall quality-of-life outcomes pre-operatively and at 6- and 12-months post-surgery using validated questionnaires. | University of Washing Quality of life questionnaire distributed pre-operatively, 6 months and 12 months.
  For the prospective cohort assess the overall quality-of-life outcomes at pre-operatively and at 6- and 12-months post-surgery using validated University of Washington Quality of Life questionnaire.
For the prospective cohort assess the swallow-related quality-of-life outcomes at pre-operatively and at 6- and 12-months post-surgery using validated questionnaires. | MD Anderson Dysphagia Inventory distributed pre-operatively, 6 months and 12 months.
  For the prospective cohort assess the swallow-related quality-of-life outcomes pre-operatively and at 6- and 12-months post-surgery using validated questionnaires.
Estimate the rates of close and involved surgical margins across all surgical salvage procedures | Through study completion, expected duration of 3 years
  Estimate the rates of close and involved surgical margins across all surgical salvage procedures
Determine the impact of close and involved margins on overall survival outcomes | Through study completion, expected duration of 3 years
  Determine the impact of close and involved margins on overall survival outcomes
Determine the impact of close and involved margins on disease-free survival outcomes | Through study completion, expected duration of 3 years
  Determine the impact of close and involved margins on disease-free survival outcomes
Determine the impact of close and involved margins on disease-specific survival outcomes | Through study completion, expected duration of 3 years
  Determine the impact of close and involved margins on disease-specific survival outcomes
Establish the rates of super-selective, selective and modified/ radical salvage neck dissection in clinically N0 and N+ necks | Through study completion, expected duration of 3 years
  Establish the rates of super-selective, selective and modified/ radical salvage neck dissection in clinically N0 and N+ necks
Ascertain how the extent of salvage neck dissection influences overall survival outcomes. | Through study completion, expected duration of 3 years
  Ascertain how the extent of salvage neck dissection influences overall survival outcomes.
Ascertain how the extent of salvage neck dissection influences disease-free survival outcomes. | Through study completion, expected duration of 3 years
  Ascertain how the extent of salvage neck dissection influences disease-free survival outcomes.
Ascertain how the extent of salvage neck dissection influences disease-specific survival outcomes. | Through study completion, expected duration of 3 years
  Ascertain how the extent of salvage neck dissection influences disease-specific survival outcomes.
Estimate the rate of occult nodal metastasis in clinically N0 necks with locally recurrent disease | Through study completion, expected duration of 3 years
  Estimate the rate of occult nodal metastasis in clinically N0 necks with locally recurrent disease
Describe the impact of neck dissection on overall survival outcomes in patients with clinically N0 necks with and without subsequent occult nodal disease | Through study completion, expected duration of 3 years
  Describe the impact of neck dissection on overall survival outcomes in patients with clinically N0 necks with and without subsequent occult nodal disease
Describe the impact of neck dissection on disease-free survival outcomes in patients with clinically N0 necks with and without subsequent occult nodal disease | Through study completion, expected duration of 3 years
  Describe the impact of neck dissection on disease-free survival outcomes in patients with clinically N0 necks with and without subsequent occult nodal disease
Describe the impact of neck dissection on disease-specific survival outcomes in patients with clinically N0 necks with and without subsequent occult nodal disease | Through study completion, expected duration of 3 years
  Describe the impact of neck dissection on disease-specific survival outcomes in patients with clinically N0 necks with and without subsequent occult nodal disease
Using multi-variate analysis, establish the clinical prognostic indicators of overall, disease free and disease specific survival. | Through study completion, expected duration of 3 years
  Establish the clinical prognostic indicators of positive survival and functional outcomes
Using multi-variate analysis, establish the clinical prognostic indicators 12 month tracheostomy and gastrostomy dependence. | Through study completion, expected duration of 3 years
  Establish the clinical prognostic indicators of functional outcomes
Compare the DNA genetic and epigenetic changes in residual, recurrent, and new primary head and neck squamous cell carcinoma with primary tumour and germline DNA samples. | Through study completion, expected duration of 3 years
  Assess the molecular makeup of head and neck tumours that have not responded to radiotherapy treatment, or which recur having previously responded.

CONTACTS AND LOCATIONS:
Overall Officials: Vinidh Paleri, Principal Investigator — Royal Marsden Hospital NHS Foundation Trust
Locations (9):
- United Kingdom (9):
  - University Hospitals Derby and Burton, Derby
  - NHS Lothian, Edinburgh
  - Western General, Greater Glasgow and Clyde, Glasgow
  - Aintree Hospital, Liverpool
  - Head and Neck Unit, Royal Marsden Hospital, London
  - Northwick Park, London
  - Oxford University Hospital NHS Foundation Trust, Oxford
  - Poole Hospital, University Hospitals Dorset, Poole
  - South Tyneside and Sunderland NHS Foundation Trust, Sunderland

IPD SHARING:
Plan to Share IPD: No